CLINICAL TRIAL: NCT02370017
Title: Combined Effect of Autologous Ex-vivo Expanded Activated NK Cell-lymphocytes (ANKL) and Doublet Chemotherapy in Patients With Advanced NSCLC as the 1st Line Treatment; Phase II
Brief Title: Combined Effect of Natural Killer Cell and Doublet Chemotherapy in Advanced NSCLC as the 1st Line Treatment
Acronym: ANKL-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Suk Young Park, M.D.-Ph.D., Professor, Medical Oncology, Dept of Internal Medicine, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUMC-ANKL-002
Record Dates: First submitted 2015-02-01; First posted 2015-02-24 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Autologous Ex vivo-expanded NK cell enriched lymphocytes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ANKL combined with chemotherapy (Experimental): combination of ANKL and doublet chemotherapy as 3rd and 4th course in patients who get stable response after initial x2 courses
  Interventions: Biological: ANKL(Ex vivo-expanded NK cell enriched lymphocytes)

INTERVENTIONS:
Biological: ANKL(Ex vivo-expanded NK cell enriched lymphocytes) — add ANKL in 3rd and 4th course in case of stable response after two initial courses

SUMMARY:
The object of this study is to identify the combined effect of ANKL and doublet chemotherapy in advanced NSCLC. The investigators design the combination of ANKL and approved chemotherapy as the 3rd and 4th courses in the patients who get stable response after x2 induction as the first line chemotherapy. ANKL (2x10*9) from peripheral blood 32ml is administered rapidly iv 12-36hr after each chemotherapeutic agents while peak effect of NK cell ligand modulation by chemotherapeutic agent is maintained. After 4th course, response evaluation is done by Response Evaluation Criteria in Solid Tumors (RECIST) and 40% or more partial response (PR, increased by 15% or more from historical control 25%) is the expected target and Simon's two stage design will be applied through the study (power 80%, a= 0.95, N1= 33, N= 68)

DETAILED DESCRIPTION:
Based on additive or synergistic effect of natural killer (NK) cell and chemotherapy (modulating the expression of NK stimulatory ligand on tumor cell), the investigators performed phase II trial of docetaxel and ANKL combination s the second line treatment in advanced non-small cell lung cancer (NSCLN) and reported the results in May 2013. (Anticancer Research 33;2115, Poster Presentation in ASCO).In that study, the investigators observed the feasibility and safety of ANKL combined with docetaxel in patients with advanced NSCLC, but the clinical benefit was not evaluated properly because the study was interrupted unintentionally and most of the enrolled patients were far advanced with large tumor burden, that is, poor immunological environment for ANKL to work.

The object of this study is to identify the combined effect of ANKL and doublet chemotherapy in advanced NSCLC. The approved doublet chemotherapy based on platinum is widely used with the response rate (RR) 25-35% after 4-6 courses as the first line treatment. The investigators design the combination of ANKL and chemotherapy as the 3rd and 4th courses in the patients who show stable response after x2 courses. Higher RR with the combination treatment is the primary outcome as compared with the chemotherapy alone - historical control; about 12% PR and 50% stable response after x2 initial courses and 25% PR after x2 more courses among the patients who get stable response after x2 initial courses. Peripheral blood 32 ml will be drawn from the patients who decide to be enrolled and about 2 weeks later ANKL (2x10*9) are scheduled to be administered rapidly iv 12-36hr after each chemotherapeutic agents while peak effect of NK cell ligand modulation by chemotherapeutic agent is maintained. After 4th course, response evaluation is done by RECIST and 40% or more PR (increased by 15% or more from historical control 25%) is the expected target and Simon's two stage design will be applied through the study (power 80%, a= 0.95, N1= 33, N= 68)

ELIGIBILITY:
Inclusion Criteria:

* advanced NSCLC with measurable lesions,
* age of 20 - 75 years, Eastern Cooperative Oncology Group (ECOG)
* performance status (PS) of 0 to 2, and stable response after x2 induction chemotherapy as first line treatment.
* No major organ dysfunction.

Exclusion Criteria:

* pregnant or lactating woman,
* active hepatitis B or C,
* AIDS or positivity for HIV, autoimmune diseases or treatment with immunosuppressive drugs,
* prior radiotherapy to the target region

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-08 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
response rate | 1 month later after 4th course
  confirmed response rate by CT scan

SECONDARY OUTCOMES:
progression free survival | 6 months
  CT or other imaging modality

CONTACTS AND LOCATIONS:
Overall Officials: Suk Young Park, MD, PhD, Principal Investigator — The Catholic University of Korea; Hoon Kim, MD, PhD, Study Director — The Catholic University of Korea
Locations (1):
- Daejeon St. Mary's Hospital, Jung-gu, Daejeon, South Korea